CLINICAL TRIAL: NCT06538207
Title: An Open-label, Uncontrolled Study of ONO-4578 and ONO-4538 in Combination With Standard-of-care Modified FOLFIRINOX (mFFX) or Gemcitabine Plus Nab-paclitaxel (GnP) Therapy as First-line Treatment in Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4578-04; jRCT2031200286 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-07-29; First posted 2024-08-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Nivolumab; Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONO-4578+ONO-4538+mFFX (Experimental)
  Interventions: Drug: ONO-4578; Drug: ONO-4538; Drug: Oxaliplatin; Drug: Levofolinate; Drug: Irinotecan; Drug: Fluorouracil
- ONO-4578+ONO-4538+GnP (Experimental)
  Interventions: Drug: ONO-4578; Drug: ONO-4538; Drug: Gemcitabine; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: ONO-4578 — Specified dose on specified days
Drug: ONO-4538 — Specified dose on specified days
  Other Names: Nivolumab
Drug: Oxaliplatin — Specified dose on specified days
  Arms: ONO-4578+ONO-4538+mFFX
Drug: Levofolinate — Specified dose on specified days
  Arms: ONO-4578+ONO-4538+mFFX
Drug: Irinotecan — Specified dose on specified days
  Arms: ONO-4578+ONO-4538+mFFX
Drug: Fluorouracil — Specified dose on specified days
  Arms: ONO-4578+ONO-4538+mFFX
Drug: Gemcitabine — Specified dose on specified days
  Arms: ONO-4578+ONO-4538+GnP
Drug: Nab-Paclitaxel — Specified dose on specified days
  Arms: ONO-4578+ONO-4538+GnP

SUMMARY:
This study is a multicenter, open-label, uncontrolled study to investigate the tolerability and safety of ONO-4578, ONO-4538, and standard of care in combination as first-line treatment in patients with metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pancreatic invasive ducatal adenocarcinoma
* 2. Life expectancy of at least 3 months
* 3. Patients with ECOG performance status 0 or 1

Exclusion Criteria:

* 1. Patients with severe complication
* 2. Patients with multiple primary cancers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities（DLT） | 28 days
Adverse event(AE) | UP to 28 days after the last dose

SECONDARY OUTCOMES:
Pharmacokinetics (Plasma concentration for ONO-4578) | Up to 28 days after the last dose
Pharmacokinetics (Serum concentration for ONO-4538) | Up to 28 days after the last dose
Overall response rate (ORR) | Up to 2 years
Disease control rate (DCR) | Up to 2 years
Overall survival (OS) | Up to 2 years
Progression-free survival (PFS) | Up to 2 years
Duration of response (DOR) | Up to 2 years
Time to response (TTR) | Up to 2 years
Best overall response (BOR) | Up to 2 years
Percentage of change in the sum of tumor diameters of target lesions | Up to 2 years
Maximum percentage of change in the sum of tumor diameters of target lesions | Up to 2 years
Changes in tumor markers (CEA and CA19-9) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (9):
- Japan (9):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Juntendo University Hospital, Bunkyō-Ku, Tokyo
  - The University of Tokyo Hospital, Bunkyō-Ku, Tokyo
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-Ku, Tokyo
  - Kyorin University Hospital, Mitaka-shi, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No